CLINICAL TRIAL: NCT03528876
Title: FOLFIRI Alternate With FOLFOX in Untreated Metastatic Gastric and Esophageal Adenocarcinoma. The LOGIC Study
Brief Title: FOLFIRI Alternate With FOLFOX in Untreated Metastatic Gastric and Esophageal Adenocarcinoma
Acronym: LOGIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Combination of chemotherapy and Immunotherapy is a new Standard of care
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Shahid Ahmed, MD, University of Saskatchewan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99183
Record Dates: First submitted 2018-05-01; First posted 2018-05-18 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Gastro-esophageal Adenocarcinoma
Keywords: gastric cancer; esophageal cancer; adnocarcinoma; FOLFIRI; FOLFOX; Metastatic cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm intervention study (Other): Biweekly FOLFOX for two cycles alternating with FOLFIRI for two cycles (FOLFOX-FOLFIRI)
  Interventions: Drug: FOLFOX and FOLFIRI

INTERVENTIONS:
Drug: FOLFOX and FOLFIRI — a biweekly regimen comprised of two cycles of FOLFOX alternating with two cycles of FOLFIRI.

SUMMARY:
Background: Gastro-esophageal (GE) cancers are a highly aggressive disease and are one of the major causes of cancer-related death worldwide. In general, combination chemotherapy has been associated with better outcomes compared with single agent chemotherapy. Fluoropyrimidine doublets FOLFOX (infusional 5FU and oxaliplatin) or FOLFIRI (infusional 5FU and irinotecan) are some of the standard first-line regimens and are less toxic than the anthracycline containing three drug regimen. Although platinum compounds are very effective in GE cancers, patients who are treated with platinum-based therapy often develop severe neuropathy and may not be able to tolerate a salvage second-line paclitaxel-based therapy.

Objectives: To evaluate progression free survival, time to progression, overall survival, toxicity and quality of life in previously untreated patients with metastatic GE cancers who will be treated with a novel biweekly regimen comprised of two cycles of FOLFOX alternating with two cycles of FOLFIRI. To determine the correlation between various clinical and pathological biomarkers including an early FDG-PET scan response and patient outcomes.

Design: Phase 2 clinical trial Methods: Thirty-six adult patients with histologically proven HER2 negative metastatic adenocarcinomas or poorly differentiated GE cancers will be recruited at the two major cancer centers in Saskatchewan over a period of two years. Patients will receive chemotherapy every two weeks and will undergo periodic imaging studies every 8 weeks. A Cox proportional analysis will be performed to assess various clinical and pathologic factors including an early FDG-PET/CT response and their correlation with patient outcomes.

Significance: The LOGIC study aims to develop an effective but potentially less toxic regimen in the management of metastatic GE cancers, offering the possibility of longer disease control as a result of 100% exposure to two active doublets in a first-line treatment setting with lower neurotoxicities and an improved rate of salvage second-line therapy. This study will inform the care of patients with metastatic GE cancers and will be used to design a larger phase 3 trial to establish a more effective but less toxic chemotherapy regimen for patients with metastatic GE cancer and to establish role of FDG-PET/CT scan and other biomarkers in predicting outcomes.

DETAILED DESCRIPTION:
1. Current Knowledge and Rationale Gastro-esophageal (GE) cancers are a highly aggressive disease and are one of the major causes of cancer-related death in the world. Despite improvements in surgical and radiation techniques and the availability of newer agents, the prognosis of recurrent GE cancers remains very poor (1-4). GE cancers comprise one of the solid organ cancers with a high fatality rate. Although 5,600 (2.8%) of the estimated 196,900 newly diagnosed cancers in Canada in 2015 were GE cancer, 4,100 (5.2%) of the 78,000 cancer related deaths were from GE cancers (3). The need for novel strategies to improve current therapy is therefore vital in the management of GE cancer.

   In many clinical trials, the treatment of metastatic gastric and esophageal cancers has merged, and the majority of patients with gastric, esophageal, or GE cancers are treated with a parallel chemotherapeutic regimens. The goal of treatment in patients with metastatic GE cancer is to control the disease, to maintain or improve quality of life, and to prolong survival. In a meta-analysis of three trials comparing chemotherapy versus best supportive care, there was a significant benefit in overall survival in favor of chemotherapy (hazard ratio [HR] 0.37; 95% CI 0.24 -0.55) (5). Hence, chemotherapy should be considered for patients with appropriate performance status.

   In general combination chemotherapy has been associated with higher response rates, and better progression free survival (PFS), and overall survival (OS) compared with single agent chemotherapy. For most patients with GE cancers combination chemotherapy represents the standard of care.

   The ECF (epirubicin, cisplatin, 5-fluorouracil) remains one of the reference regimens for the first-line treatment of metastatic GE cancers. However, when both oxaliplatin (O) and capecitabine (X) are substituted for cisplatin (C) and 5FU (F), respectively in the ECF regimen (EOX, EOF, ECX), outcomes are at least as good as with ECF (6). FOLFOX has also been compared to ECF with comparable results. An intergroup phase 2 trial evaluated ECF, irinotecan and cisplatin (IC), or FOLFOX in combination with cetuximab, and concluded that response rates, PFS, and median OS were comparable in the ECF and FOLFOX groups. FOLFOX-based regimen required fewer treatment modifications compared with other regimens (7).

   Irinotecan-based regimens also appeared to be superior to cisplatin/5FU in response rates and survival being in the 10-12 month range (8,9). A randomized phase 3 trial evaluated 416 patients with advanced gastric or esophagogastric junction (EGJ) adenocarcinoma who were assigned to either FOLFIRI or ECX (10). There were no significant differences in median PFS, OS, or response rates between the two regimens. Time to treatment failure favored FOLFIRI (5.1 versus 4.2 months). Furthermore, FOLFIRI was better tolerated overall (rate of grade 3 or 4 toxicity 69 versus 84% with ECX). Although docetaxel based regimens such as DCF have shown significant improvement in response, PFS, and OS compared to cisplatin/5-FU, it is a more toxic regimen with a higher rates of grade 3 or 4 toxicities and is not commonly used in Canada (11-13).

   Despite a large number of randomized trials, there is no globally accepted, standard first-line chemotherapy regimen in advanced HER2 negative GE cancer. A meta-analysis of first-line chemotherapy trials for metastatic GE cancers involving 10,249 patients in 50 trials that incorporated 17 different chemotherapy regimens with 37 direct comparisons showed that anthracycline-containing triplets such as ECF or EOX and the docetaxel-containing triplet DCF were more toxic but not superior to fluoropyrimidine doublets with respect to PFS or OS (14). Although fluoropyrimidine noncisplatin-containing doublets, fluoropyrimidine-cisplatin doublets, and all triplet regimens showed significant improvements in overall survival compared with fluoropyrimidine alone, a fluoropyrimidine-noncisplatin doublet containing oxaliplatin (FOx) or irinotecan (FI) significantly improved OS compared with a fluoropyrimidine plus cisplatin doublet (for FI, the HR for death was 0.85, 95% CI 0.71-0.99; for FOx, the HR was 0.83, 95% CI 0.71-0.98). The cisplatin/fluoropyrimidine doublet was also associated with more grade 3 or 4 toxicity. Furthermore, an individual patient data meta-analysis of the GASTRIC group involving 4245 patients of 55 eligible trials concluded that there was no role for epirubicin in combination with a fluoropyrimidine and a platinum agent (15).

   Hence, based on efficacy and toxicity profiles, fluoropyrimidine doublets FOLFOX or FOLFIRI are the preferred first-line therapy over cisplatin doublets, anthracycline triplets, and DCF. A substantial number of patients who have disease progression after a first-line chemotherapy may not undergo further active therapy, mainly because of deterioration of their performance status or side effects-related to previous treatments. Although the combinations of 5-FU with irinotecan and oxaliplatin (FOLFOXIRI) is an active regimen in colorectal and pancreatic cancer, it has been associated with a higher rate of adverse effects. Furthermore, this regimen is currently administered at the two major treatment centers in Saskatchewan requiring frequent long-distance travel.

   The LOGIC study aims to evaluate efficacy and toxicity of a novel regimen comprised of biweekly FOLFOX for two cycles alternating with FOLFIRI for two cycles (FOLFOX-FOLFIRI) as the first-line therapy for patients with previously untreated metastatic GE cancers. This novel schedule will expose the patients to three active agents in the first-line setting without the toxicity that is typically associated when all of three drugs are given together. Furthermore, since oxaliplatin is associated with significant neuropathy, decreasing the exposure of this drug in an alternating schedule can result in less cumulative neurotoxicity and an increased use of second-line treatment.
2. Research Questions and Hypothesis

   * Whether a novel treatment regimen comprised of biweekly FOLFOX alternating with FOLFIRI as a first-line therapy for patients with previously untreated metastatic GE cancers is as effective and less toxic compared to the other available two- and three-drug regimens?
   * Whether an early fluorodeoxyglucose-positron emission tomography (FDG-PET) scan response and other biomarkers correlate with better PFS and OS in patients with metastatic GE cancer who are treated with FOLFOX alternating with FOLFIRI?
   * What is rate of second-line therapy in patients with metastatic GE cancer who received first-line FOLFOX alternating with FOLFIRI?
   * We hypothesize that this novel regimen FOLFOX-FOLFIRI is less toxic but at least as effective as the other two- and three-drug regimens available in metastatic GE cancer and that an early FDG-PET response is associate with a better PFS rate. We also hypothesize that this novel regimen is associated with low rate of decline in QOL at 3 and 6 months.
3. Objectives

   3.1 Primary Objectives
   * To evaluate progression-free survival of patients with metastatic GE cancer who are treated with FOLFOX-FOLFIRI.
   * To determine correlation between various clinical and pathological biomarkers including an early FDG-PET scan response and progression free survival and QOL of patients who are treated with FOLFOX-FOLFIRI.

   3.2 Secondary Objectives
   * To assess the quality of life of patients who are treated with FOLFOX alternating with FOLFIRI.
   * To determine the response rate, time to treatment failure, and overall survival of patients who are treated with FOLFOX alternating with FOLFIRI.
   * To evaluate treatment toxicities, including the rate of neurotoxicity with FOLFOX alternating with FOLFIRI.
4. Eligibility Criteria 4.1 Inclusion Criteria

   * Adult patients (≥18 years older) with histologically proven HER2 negative adenocarcinoma or poorly differentiated carcinoma of the esophagus, GE junction tumors, and gastric cancer.
   * Measurable or assessable metastatic disease.
   * Performance status World Health Organization (WHO) 0-2 and life expectancy of greater than 3 months.
   * No previous chemotherapy for advanced disease.
   * Adequate functioning of the bone marrow, liver, and kidneys. 4.2 Exclusion Criteria
   * Breastfeeding or pregnancy.
   * Active second primary cancer except in situ cancer or non-melanoma skin cancer.
   * Cerebral metastases or leptomeningeal carcinomatosis.
   * Severe or uncompensated concomitant medical conditions including peripheral neuropathy.
5. Methods

   5.1 Study design
   * The LOGIC trial is a single arm phase 2 study. 5.2 Sample size
   * Based on response rates of 40-50% with combination chemotherapy in the randomized trials, to achieve 80% power the required sample in this single arm study is N=36 with 5% significance level and two-sided test. At this power we will be able to do appropriate analyses and meaningful comparison of efficacy and toxicity.

   5.3 Recruitment timeline

   • Each year approximately 100 patients are diagnosed with gastric, esophageal, and gastro-esophageal cancer in Saskatchewan. Unfortunately, most patients either have advanced disease at diagnosis or develop recurrent cancer after curative treatment. Based on that we estimated that each month we will be able to recruit 2 to 3 patients at the two major cancer centers (the Saskatoon Cancer Center and the Allan Blair Cancer Center) in Saskatchewan and recruitment will be completed in 18-24 months.

   5.4 Analysis

   • Response rates and stable disease rates will be summarized by percentages and their 95% CI. Survival curves will be analyzed using the Kaplan-Meier method, and differences between groups will be analyzed using log-rank test. The efficacy and toxicities of this novel regime will be compared with the historical control from the publish literature. Correlation will be significant at the 0.05 level (two tailed). Univariate analyses will be done to assess various clinical and pathologic factors for their correlation with prognosis and if feasible a multivariate analysis will be performed. Linear mixed models will be used to assess changes over time for overall QOL and for separate components of QOL.
6. Chemotherapy Regimen

   6.1 FOLFOX Drug Dosage Timing Oxaliplatin 85 mg/m2 Day 1 Leucovorin 400 mg/m2 Day 1 Fluorouracil 400 mg/m2 Day 1 Fluorouracil 2400 mg/m2 48 hrs infusion
   * for patients with ECOG P 6.2 FOLFIRI Drug Dosage Timing Irinotican 180 mg/m2 Day 1 Leucovorin 400 mg/m2 Day 1 Fluorouracil 400 mg/m2 Day 1 Fluorouracil 2400 mg/m 48 hrs infusion
   * for patients with ECOG P
7. Assessment, interventions, and follow-up visits 7.1 Baseline Assessment

   * Pretreatment patient evaluation includes a complete clinical history and physical examination, full blood counts, renal and liver function tests (bilirubin, AST, alkaline phosphatase), albumin, electrolytes, magnesium, calcium, serum carcinoembryonic (CEA) level measurements, and CT scan of the thorax, abdomen, and pelvis (a baseline scan within 4 weeks of start of treatment, and then with every 4th cycles).
   * Responses will be evaluated with standard Response Evaluation Criteria in Solid Tumors (RECIST) by means of CT scans and will be complemented by an FDG-PET/CT scan.

   7.2 Follow-up visits

   • Patients will be seen prior to the second cycle of FOLFOX and FOLFIRI and before every other infusion with medical history, examination and CBC and differential, platelets, creatinine, LFT's (bilirubin, AST, alkaline phosphatase), electrolytes, albumin, and blood Pressure measurement.

   7.3 Dose Modification
   * Toxicity will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria Version 4.
   * Specific drug reductions and management of neurotoxicity will be made in accordance with published recommendations for FOLFOX and FOLFIRI at the discretion of treating oncologist.

   7.4 Response Assessment

   • Responses will be evaluated with standard Response Evaluation Criteria in Solid Tumors (RECIST) by means of CT scans and will be complemented by an FDG-PET/CT scan.

   7.5 Treatment Duration A maximum of 12 cycles is planned, but treatment could be continued off the protocol in patients without disease progression in cases of clinical benefit. Second-line chemotherapy will be left to the discretion of the treating physician.
8. Quality of Life

   * Quality of life (QOL) focuses on patient construct. Physical health, functional status, sexual, and psychosocial domains are considered key elements in QOL measurement. The European Organization for Research and the Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) along with the EORTC Esophago-Gastric Cancer Module (QLQ-OG25).
   * The EORTC QLQ-C30 is a widely used instrument for measuring general cancer QOL. It consists of 30 items and patients responses are transformed to produce 0-100 scores on five functional scales, nine symptom scales and a scale representing global quality of life. Higher functional scale scores indicate better QOL whereas higher symptom scale/item scores indicate higher level of symptoms.
   * The QLQ-OG25 has six scales, dysphagia, eating restrictions, reflux, odynophagia, pain and anxiety. The QLQ-OG25 is recommended to supplement the EORTC QLQ-C30 when assessing HRQL in patients with esophageal, junctional or gastric cancer (16). Both English and French versions of questionnaire are available. The QOL will be measured at baseline and then every four weeks till disease progression.
9. Correlative science

   * Positron Emission Tomography is commonly used to complement anatomic imaging in cancer management (17). A CT-PET scan allows for images representing both anatomic and metabolic properties. A PET/CT has emerged as an effective tool for diagnostic and therapeutic evaluation in many types of cancers, including GE cancers. Evidence has suggested that FDG-PET/CT seems to be an effective noninvasive tool for response assessment in GE cancer (18,19). Early FDG-PET response will be correlated with PFS and QOL.
   * In addition, the correlation between outcomes and various biomarkers such as tumor grade, lymphocyte to neutrophil ratio, E-cadherin, fibroblast growth factor receptor, TP53, and microsatellite instability will be evaluated. Immunohistochemical analysis of paraffin embedded tumor specimens using antibodies against several biomarkers including P53, MLH1, MSH2, MSH6, PMS2, E-cadherin, fibroblast growth factor receptor, and Ki-67 will be performed. In addition, we will use the plasma proteome database (http://www.plasmaproteomedatabase.org) to identify novel biomarkers. The purpose of these analyses is to identify differentially expressed tumor-specific genes that code for the plasma proteome.
   * We will select tumor markers based on their gradient of differential expression and examine at least four markers using ELISA assays in patient's plasma samples (at 0 and 2 months of treatment) to assess their predictive and prognostic values.
10. Significance

    * Based on the indirect evidence that anthracycline-containing triplets such as ECF or EOX or docetaxel-containing triplets such as DCF are more toxic but not superior to fluoropyrimidine doublets such as FOLFOX or FOLFIRI, this study aims to develop an effective novel but potentially less toxic regimen in the management of metastatic GE cancers, offering the possibility of longer disease control as a result of 100% exposure to two active doublets in a first-line treatment setting and an improvement in the rate of salvage second line therapy.
    * Furthermore, this study will evaluate an early FDG-PET/CT response and various other clinical and pathological variables and their correlation with PFS and QOL using this novel regimen with an ultimate goal to improve care of this highly fatal cancer. The results will be used for future collaboration and development of a late phase trial at the national level.
11. Knowledge Translation

    * The research findings will be presented to health professionals, patients and their family and decision makers using various platform. The findings will be shared with P & T committee and PFAC members. The result will be presented to the Western Canadian Gastrointestinal Cancer groups. The findings will be published in the peer reviewed scientific journals and will be presented at international, national and local conferences.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years older) with histologically proven HER2 negative adenocarcinoma or poorly differentiated carcinoma of the esophagus, GE junction tumors, and gastric cancer.
* Measurable or assessable metastatic disease.
* Performance status World Health Organization (WHO) 0-2 and life expectancy of greater than 3 months.
* No previous chemotherapy for advanced disease.
* Adequate functioning of the bone marrow, liver, and kidneys.

Exclusion Criteria:

* Breastfeeding or pregnancy.
* Active second primary cancer except in situ cancer or non-melanoma skin cancer.
* Cerebral metastases or leptomeningeal carcinomatosis.
* Severe or uncompensated concomitant medical conditions including peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Progression free survival | At 12 months
  Time from enrollment till the date of disease progression

SECONDARY OUTCOMES:
overall survival | At 3 years
  Time from enrollment till death from any cause
Metabolic response rate | At 2 months
  change in baseline SUV of PET-CT after 4 cycles of chemotherapy
Neurotpathy | At 6 and 12 months
  grade 3/4 neuropathy
Decline in quality of life | At 6 and 12 months
  The European Organization for Research and the Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30) along with the EORTC Esophago-Gastric Cancer Module (QLQ-OG25).

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Ahmed, Md, PhD, Principal Investigator — University of Saskatchewan
Locations (2):
- Canada (2):
  - Allan Blair Cancer Center, Regina, Saskatchewan
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No